CLINICAL TRIAL: NCT00185536
Title: Effects of Advertising on Young Children's Perception of Taste
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Other Study IDs: 80618; 20664
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Obesity
Keywords: Taste; preschool children; fast food
MeSH Terms: conditions — Obesity | interventions — Product Packaging

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Packaging and identification of source

SUMMARY:
To test whether young children's actual taste preferences are influenced by the natural marketing environment in which they live. To do so, we tested whether preschool children would like the taste of a food more if they thought it was from a heavily marketed source. We asked preschool children to taste identical foods in packaging from this heavily marketed source and plain packaging, and to tell us if they tasted the same or if one tasted better. We hypothesized that, even among a sample of 3-5 year olds participating in Head Start, a federally-sponsored preschool program for low-income families, young children would prefer the taste of foods perceived to be from the heavily marketed source.

ELIGIBILITY:
Inclusion Criteria:

* enrolled at participating head start sites

Exclusion Criteria:

* unable to complete the study procedures

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-04

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N. Robinson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Robinson TN, Borzekowski DL, Matheson DM, Kraemer HC. Effects of fast food branding on young children's taste preferences. Arch Pediatr Adolesc Med. 2007 Aug;161(8):792-7. doi: 10.1001/archpedi.161.8.792. PMID 17679662